CLINICAL TRIAL: NCT04919681
Title: Efficacy of a Stretching Protocol on Regional and Distant Pain Sensitivity:
Brief Title: Efficacy of Stretching on Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other); Research Unit for General Practice in Aalborg (Other)
Responsible Party: Principal Investigator, Morten Pallisgaard, Associate Lecturer, University College of Northern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UniversityCND3
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Pain Threshold
Keywords: Stretching; Pain sensitivity; Range of motion; Exercise adherence
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Single-blind longitudinal repeated measures study
Masking Description: Participants are blinded to the results of the pressure pain threshold measurements. Participants and examiner are blinded to the results of the range of motion and passive resistive torque measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stretching (Experimental): Static stretching of the knee flexors
  Interventions: Other: Stretch exercises

INTERVENTIONS:
Other: Stretch exercises — The intervention comprises of six weeks daily bi-lateral static stretching of the knee flexors. Stretches are performed seated on the ground. The participant sits upright on the floor with one leg straight. The sole of the other foot should be placed on the inside of the outstretched leg. The participant leans slightly forward, trying to touch their toes while maintaining full knee extension. Stretching is performed to the point of discomfort, and each stretch is held for 30-seconds for three repetitions.

SUMMARY:
The primary objective of this study is to determine the immediate efficiency of a six weeks regular stretching protocol on regional and distant pain sensitivity. It is hypothesised that regional and distant pain sensitivity will significantly decrease following six weeks of regular stretching.

The secondary objective of the study is to determine the effect after four-week cessation of the stretching protocol on regional and distant pain sensitivity. If regional and distant pain sensitivity decrease following regular stretching, it is hypothesised that the analgesic effect will abate following four-week cessation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-65 years are recruited. As part of the screening, volunteers will also be asked to indicate known medical issues or diseases. Participants are included if they have no known medical conditions such as
* cognitive impairments,
* neurological,
* orthopaedic,
* or neuromuscular problems that might affect the somatosensory system or preclude stretching exercises or range of motion testing at the knee.

Exclusion Criteria:

* Individuals who regularly engage in flexibility training (e.g., stretching, tai chi, pilates or yoga)
* or use any medication that might affect the somatosensory system, such as pain medication, are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity | Baseline
  The primary outcome is pain sensitivity expressed as regional and distant pressure pain thresholds measured by a handheld pressure algometer
Pain sensitivity | 6 weeks
  The primary outcome is pain sensitivity expressed as regional and distant pressure pain thresholds measured by a handheld pressure algometer
Pain sensitivity | 10 weeks
  The primary outcome is pain sensitivity expressed as regional and distant pressure pain thresholds measured by a handheld pressure algometer

SECONDARY OUTCOMES:
Range of motion | Baseline
  Passive knee extension range of motion measured by the Biodex system 4 pro isokinetic dynamometer
Range of motion | 6 weeks
  Passive knee extension range of motion measured by the Biodex system 4 pro isokinetic dynamometer
Range of motion | 10 weeks
  Passive knee extension range of motion measured by the Biodex system 4 pro isokinetic dynamometer
Passive resistive torque | Baseline
  Passive resistive torque measured in passive kne extension measured by the Biodex system 4 pro isokinetic dynamometer
Passive resistive torque | 6 weeks
  Passive resistive torque measured in passive kne extension measured by the Biodex system 4 pro isokinetic dynamometer
Passive resistive torque | 10 weeks
  Passive resistive torque measured in passive kne extension measured by the Biodex system 4 pro isokinetic dynamometer

OTHER OUTCOMES:
Adherence to the stretching protocol | 6 weeks
  Adherence to the stretching protocol will be measured using self-reported data from an mHealth app.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachmann, Msc., Study Director — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data is made available upon request.
Supporting Information: Study Protocol
Time Frame: Study protocol will be published
Access Criteria: The study protocol will be published open access

REFERENCES:
- [Derived] Stove MP, Thomsen JL, Magnusson SP, Riis A. The effect of six-week regular stretching exercises on regional and distant pain sensitivity: an experimental longitudinal study on healthy adults. BMC Sports Sci Med Rehabil. 2024 Sep 27;16(1):202. doi: 10.1186/s13102-024-00995-2. PMID 39334218